CLINICAL TRIAL: NCT02655302
Title: Study of the Involvement of IL-17 / IL-22 Pathway in Bacterial Exacerbations of COPD
Acronym: COPD1722
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2013_76; 2015-A00190-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2015-12-03; First posted 2016-01-14 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Bacterial Infections
Keywords: Interleukin-17; Interleukin-22; Microbiota; Exacerbations; Immunity; Mucosal
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bacterial exacerbations (Other): Patients with at least 10^7 UFC/ml bacteria in their sputum during their first COPD exacerbation.
  Interventions: Other: Sample collecting; Other: Lung function measure
- Non-bacterial exacerbations (Other): Patients without detected bacteria or below 10^7 UFC/ml in sputum during their first COPD exacerbation.
  Interventions: Other: Sample collecting; Other: Lung function measure

INTERVENTIONS:
Other: Sample collecting — Collect sputum, blood and nasopharyngeal swab during the exacerbation and at steady state 8 to 16 weeks later.
Other: Lung function measure — Measure lung function and follow it during 4 years

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a worldwide chronic inflammatory disease of the airways linked to environmental exposure. The chronic course of COPD is often interrupted by acute exacerbations which have a major impact on the morbidity and mortality of COPD patients. A bacterial etiology for these exacerbations is common (almost 50%). Moreover, airway bacterial colonization linked to an increased susceptibility is observed in COPD patients. Effective Th17 immune response is needed to develop a good response against bacteria. Thus, this study aims to demonstrate that there is a defective IL-17/ IL-22 response to bacteria in COPD leading to airway bacterial colonization and infection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed COPD according GOLD guidelines
* Current or ex-smoker (at least 10 pack-years)
* Hospitalized for COPD exacerbation

Exclusion Criteria:

* Asthma or Cystic fibrosis
* No other chronic lung disease
* Solid Tumor unhealed or not considered in remission
* Inhaled drug consumption
* Women of childbearing potential without effective contraception
* Pregnant or breastfeeding women
* Incapable of consent
* Lack of social security coverage

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-04 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Measure cytokines by ELISA | At inclusion (exacerbation) and between 8 to 16 weeks (steady-state)
  Compare the delta of IL-17 and IL-22 cytokines between exacerbation and steady-state in the sputum,between the two groups of patients.

SECONDARY OUTCOMES:
Compare the delta of IL-17 and IL-22 cytokines between exacerbation and steady-state in the blood. | At inclusion (exacerbation) and between 8 to 16 weeks (steady-state)
  Measure cytokines by ELISA in the blood at exacerbation and at steady-state. Compare the delta of these cytokines between the two groups of patients.
Identify IL-17 and IL-22 producing cells in the blood | At inclusion (exacerbation) and between 8 to 16 weeks (steady-state)
  Identify by flow cytometry, IL-17 and/or IL-22 positive immune cell types in the blood.
Identify IL-17 and IL-22 producing cells in the sputum | At inclusion (exacerbation) and between 8 to 16 weeks (steady-state)
  Identify by flow cytometry, IL-17 and/or IL-22 positive immune cell types in the sputum.
Quantification of immune cell types in the blood | At inclusion (exacerbation) and between 8 to 16 weeks (steady-state)
  Quantify by flow cytometry different immune cells in the blood: monocytes, macrophages, B and T cells, innate lymphocytes.
Quantification of immune cell types in the sputum | At inclusion (exacerbation) and between 8 to 16 weeks (steady-state)
  Quantify by flow cytometry different immune cells in the sputum: monocytes, macrophages, B and T cells, innate lymphocytes.
Quantification of pro-inflammatory cytokines in blood | At inclusion (exacerbation) and between 8 to 16 weeks (steady-state)
  Quantify by ELISA Th1 (IL-12, IFN gamma), Th2 (IL-4, IL-5), Th17 (IL-1 beta, IL-6, IL-23, TGF beta), regulatory (IL-10) and pro-inflammatory cytokines (IL-8) in the blood.
Quantification of pro-inflammatory cytokines in sputum | At inclusion (exacerbation) and between 8 to 16 weeks (steady-state)
  Quantify by ELISA Th1 (IL-12, IFN gamma), Th2 (IL-4, IL-5), Th17 (IL-1 beta, IL-6, IL-23, TGF beta), regulatory (IL-10) and pro-inflammatory cytokines (IL-8) in the sputum.
Identify pathogens linked to the exacerbation | At inclusion (exacerbation)
  Research of classical bacteria and fungi by usual microbial cultures from sputum and of respiratory virus and non conventional bacteria (Mycoplasma, Legionella, Bordetella pertussis and parapertussis and Chlamydophila pneumoniae) by PCR on nasopharyngeal swab.
Identify persistent pathogens at steady-state | Between 8 to 16 weeks (steady-state)
  Research of classical bacteria and fungi by usual microbial cultures from sputum and of respiratory virus and non conventional bacteria (Mycoplasma, Legionella, Bordetella pertussis and parapertussis and Chlamydophila pneumoniae) by PCR on nasopharyngeal swab.
Compare sputum microbiota between exacerbation and steady-state | At inclusion (exacerbation) and between 8 to 16 weeks (steady-state)
  Metagenomic analysis on sputum
Compare oxidative stress in the blood between exacerbation and steady-state | At inclusion (exacerbation) and between 8 to 16 weeks (steady-state)
  Quantification by ELISA in the blood of oxidative stress markers (isoprostane, superoxyde dismutase, 3-nitrotyrosine, peroxyde, catalase).
Quantification of oxidative stress in exhaled condensates | At inclusion (exacerbation) and between 8 to 16 weeks (steady-state)
  Quantification by ELISA of nitrite species in exhaled condensates.
Describe exacerbation phenotype | At inclusion (exacerbation)
  Collect respiratory symptoms, received treatments and hospitalization duration.
Describe environmental exposure | At inclusion (exacerbation), between 8 to 16 weeks (steady-state) and annually for 4 years
  Collect informations on the patient's occupation, occupational exposures and smoking.
Describe COPD clinical phenotype | At inclusion (exacerbation), between 8 to 16 weeks (steady-state) and annually for 4 years
  Collect morphological informations, history of exacerbations
Describe COPD radiological phenotype | Between 8 to 16 weeks (steady-state)
  Realization of a chest CT scan if not performed during the 2 previous years.
Quantify Quality of Life | At inclusion (exacerbation), between 8 to 16 weeks (steady-state) and annually for 4 years
  Realization of the COPD Assessment Test (CAT), a quality of life questionnaire.
Describe COPD treatments | At inclusion (exacerbation), between 8 to 16 weeks (steady-state) and annually for 4 years
  Collect informations on treatments related to COPD including inhaled treatments, influenza and pneumococcal vaccinations, oxygen therapy and respiratory rehabilitation.
Measure static lung function | Between 8 to 16 weeks (steady-state) and annually for 4 years
  Test the lung function with spirometry and plethysmography repeated annually to measure the decline of respiratory function.
Measure airway resistances | Between 8 to 16 weeks (steady-state) and at 2 and 4 years
  Measure resistances with the forced oscillation technique.
Measure exercise tolerance | At inclusion (end of the hospitalization for exacerbation), between 8 to 16 weeks (steady-state) and annually for 4 years
  Perform a 6-minute walk-test.
Analysis exercise tolerance | Between 8 to 16 weeks (steady-state) and at 2 and 4 years
  Perform a cardiopulmonary exercise test on a bicycle.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Bautin, MD, Principal Investigator — University Hospital, Lille
Locations (4):
- France (4):
  - University hospital of Lille, Lille
  - Roubaix hospital, Roubaix
  - Seclin hospital, Seclin
  - Tourcoing hospital, Tourcoing

IPD SHARING:
Plan to Share IPD: No